CLINICAL TRIAL: NCT01710657
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of Lacosamide as Adjunctive Therapy in Japanese and Chinese Adults With Uncontrolled Partial-Onset Seizures With or Without Secondary Generalization
Brief Title: A Trial to Evaluate the Efficacy and Safety of Adjunctive Therapy With Lacosamide in Adults With Partial-Onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma SA (Industry)
Collaborators: UCB Japan Co. Ltd. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EP0008; 2014-003622-41 (EudraCT Number); JapicCTI-121988 (Registry Identifier: JAPIC)
Record Dates: First submitted 2012-10-17; First posted 2012-10-19 (Estimated); Results first posted 2015-02-09 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-07

CONDITIONS: Epilepsy; Partial Onset Seizures
Keywords: Lacosamide; Epilepsy; Partial Onset Seizures
MeSH Terms: conditions — Epilepsy | interventions — Lacosamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Matching placebo for 16 weeks.
  Interventions: Drug: Placebo
- Lacosamide 200 mg/day (Experimental): Lacosamide treatment of 200 mg/day (100 mg bid (twice daily)) for 16 weeks.
  Interventions: Drug: Lacosamide 50 mg; Drug: Lacosamide 100 mg
- Lacosamide 400 mg/day (Experimental): Lacosamide treatment of 400 mg/day (200 mg bid (twice daily)) for 16 weeks.
  Interventions: Drug: Lacosamide 50 mg; Drug: Lacosamide 100 mg

INTERVENTIONS:
Drug: Lacosamide 50 mg — * Active Substance: Lacosamide
  * Pharmaceutical Form: Film-coated tablet
  * Concentration: 50 mg
  * Route of Administration: Oral use
  Other Names: Vimpat
  Arms: Lacosamide 200 mg/day; Lacosamide 400 mg/day
Drug: Lacosamide 100 mg — * Active Substance: Lacosamide
  * Pharmaceutical Form: Film-coated tablet
  * Concentration: 100 mg
  * Route of Administration: Oral use
  Other Names: Vimpat
  Arms: Lacosamide 200 mg/day; Lacosamide 400 mg/day
Drug: Placebo — Matching oral Placebo tablets twice daily for 16 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of 200 and 400 mg/day of orally administered Lacosamide as adjunctive therapy compared with placebo in Japanese and Chinese adults with uncontrolled Partial-Onset Seizures with or without secondary generalization.

ELIGIBILITY:
Inclusion Criteria:

* Subject has had an Electroencephalogram (EEG) and a brain Computerized Tomography (CT) scan or Magnetic Resonance Imaging (MRI) exam consistent with a Diagnosis of Epilepsy with Partial-Onset Seizures according to the International Classification of Epileptic Seizures (1981)
* Subject must have been observed to have Partial-Onset Seizures for at least the previous 2 years despite prior therapy with at least 2 Anti-Epileptic Drugs (AEDs)(concurrently or sequentially) and must have been observed to have on average at least 4 Partial-Onset Seizures per 28 days with a seizure-free phase no longer than 21 days in the 8-Week Period prior to entry into the Baseline Period. In the case of Simple Partial Seizures, only those with motor signs will be counted towards meeting the inclusion criterion
* Subjects must be on a stable dose regimen of at least 1, but no more than 3 AEDs (concurrent stable Vagus Nerve Stimulation (VNS) is not counted as an AED). The VNS must have been in place for at least 6 months prior to study entry. The dosage of concomitant AED therapy and the settings of the VNS must be kept constant for a period of at least 4 weeks prior to entry into the Baseline Period
* Minimum Body Weight of 40 kg

Exclusion Criteria:

* Subject has a lifetime history of suicide attempt (including an active attempt, interrupted attempt, or aborted attempt) or has a suicidal ideation in the past 6 months as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening
* Subject has a current or previous diagnosis of Pseudo-Seizures, Conversion Disorders, or other non-epileptical events that could be confused with Seizures
* Subject has Seizures that are uncountable due to Clustering (ie, an episode lasting less than 30 minutes in which several Seizures occur with such frequency that the initiation and completion of each individual Seizure cannot be distinguished) during the 8-Week Period prior to Visit 1
* Subject has a history of Primary Generalized Seizures
* Subject with a history of Status Epilepticus within the 12-Months Period prior to Visit 1
* Subject who underwent surgery for Epilepsy within the 2 Years Period prior to Visit 1
* Subjects with cardiac, renal, hepatic, endocrinological dysfunction or psychiatric illness that may impair reliable participation in the study or necessitate the use of medication not allowed by the protocol

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 548 (Actual)
Dates: Start 2012-09; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (76):
- China (31):
  - 86026, Beijing
  - 86027, Beijing
  - 86015, Changchun
  - 86005, Chengdu
  - 86032, Chengdu
  - 86006, Chongqing
  - 86031, Dalian
  - 86009, Guanghzou
  - 86007, Guangzhou
  - 86008, Guangzhou
  - 86013, Guangzhou
  - 86016, Guangzhou
  - 86014, Hangzhou
  - 86010, Harbin
  - 86019, Jinan
  - 86004, Kunming
  - 86011, Nanchang
  - 86012, Nanchang
  - 86028, Nanjing
  - 86003, Qingdao
  - 86001, Shanghai
  - 86023, Shanghai
  - 86025, Shanghai
  - 86021, Shenyang
  - 86020, Shijiazhuang
  - 86022, Suzhou
  - 86002, Taiyuan
  - 86018, Wuhan
  - 86024, Wuhan
  - 86017, Xi'an
  - 86029, Xiamen
- Japan (45):
  - 81056, Asaka
  - 81030, Fujisawa
  - 81013, Fukuoka
  - 81054, Fukuoka
  - 81057, Hachinohe
  - 81008, Hakodate
  - 81027, Hamamatsu
  - 81004, Himeji
  - 81018, Hiroshima
  - 81019, Iwanuma
  - 81012, Kagoshima
  - 81033, Kitakyushu
  - 81017, Kobe
  - 81024, Kodaira
  - 81010, Kokubunji
  - 81032, Kōshi
  - 81014, Kurume
  - 81047, Kyoto
  - 81035, Nagakute
  - 81028, Nagoya
  - 81029, Nagoya
  - 81040, Nara
  - 81007, Neyagawa
  - 81002, Niigata
  - 81046, Ohmura
  - 81005, Okayama
  - 81011, Saitama
  - 81042, Sakai
  - 81025, Sapporo
  - 81048, Sapporo
  - 81053, Sapporo
  - 81009, Sayama
  - 81020, Sendai
  - 81031, Sendai
  - 81021, Shimotsuke
  - 81022, Shimotsuke
  - 81026, Shinjuku
  - 81003, Shizuoka
  - 81023, Suita
  - 81051, Suita
  - 81052, Suita
  - 81016, Takatsuki
  - 81006, Toyonaka
  - 81050, Ube
  - 81001, Yamagata

REFERENCES:
- [Result] Doty P, Hebert D, Mathy FX, Byrnes W, Zackheim J, Simontacchi K. Development of lacosamide for the treatment of partial-onset seizures. Ann N Y Acad Sci. 2013 Jul;1291(1):56-68. doi: 10.1111/nyas.12213. PMID 23859801
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 676 subjects with uncontrolled partial-onset seizures (of the 676 subjects, the number of Chinese subjects and Japanese subjects was planned to be 507 and 169, respectively) was planned to be screened and 540 subjects were planned to be enrolled in all regions of Japan and China.
Pre-assignment Details: Overall, 692 subjects were screened and 548 subjects were enrolled. The Participant Flow refers to the Safety Set (SS) which was defined as all enrolled subjects who took at least 1 dose of Lacosamide. Reasons for discontinuation were only calculated for the SS. 547 subjects were included in the Safety Set.
Groups:
- Lacosamide 200 mg/Day: Lacosamide Treatment of 200 mg/day (100 mg bid) for 16 weeks.
  Lacosamide 50 mg: - Active Substance: Lacosamide
  * Pharmaceutical Form: Film-coated tablet
  * Concentration: 50 mg
  * Route of Administration: Oral use
  Lacosamide 100 mg: - Active Substance: Lacosamide
  * Pharmaceutical Form: Film-coated tablet
  * Concentration: 100 mg
  * Route of Administration: Oral use
- Lacosamide 400 mg/Day: Lacosamide Treatment of 400 mg/day (200 mg bid) for 16 weeks.
  Lacosamide 50 mg: - Active Substance: Lacosamide
  * Pharmaceutical Form: Film-coated tablet
  * Concentration: 50 mg
  * Route of Administration: Oral use
  Lacosamide 100 mg: - Active Substance: Lacosamide
  * Pharmaceutical Form: Film-coated tablet
  * Concentration: 100 mg
  * Route of Administration: Oral use
Period: Overall Study
Arm/Group | Placebo | Lacosamide 200 mg/Day | Lacosamide 400 mg/Day
Started | 184 | 183 | 180
Titration Period (4 Weeks) | 184 | 183 | 180
Maintenance Period (12 Weeks) | 176 | 175 | 168
Completed | 166 | 171 | 148
Not Completed | 18 | 12 | 32
Not completed — Lost to Follow-up | 2 | 0 | 1
Not completed — Protocol Violation | 2 | 2 | 0
Not completed — Adverse Event | 14 | 8 | 28
Not completed — Withdrawal by Subject | 0 | 1 | 2
Not completed — Lack of Efficacy | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Baseline Characteristics refer to the Safety Set (SS) which was defined as all enrolled subjects who took at least 1 dose of Lacosamide.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lacosamide 200 mg/Day | Lacosamide 400 mg/Day | Total
Number analyzed (Participants) | 184 | 183 | 180 | 547
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 18 | 15 | 53
  Between 18 and 65 years | 164 | 163 | 164 | 491
  >=65 years | 0 | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (12.0) | 33.2 (12.2) | 32.3 (11.9) | 32.4 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 89 | 76 | 247
  Male | 102 | 94 | 104 | 300
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 184 | 183 | 180 | 547
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Chinese | 136 | 136 | 133 | 405
  Japanese | 48 | 47 | 47 | 142

OUTCOME MEASURES:

1. Primary Outcome: Change in Partial-Onset Seizure Frequency Per 28 Days From Baseline to the Maintenance Period
Description: Partial-onset seizure (POS) frequency per 28 days was calculated as:
  POS frequency = (Number of POS over the specified time interval) / (Number of days in the interval with available diary data) x 28.
  A negative value in Change in Partial-onset seizure frequency indicates a reduction of Partial-onset seizure frequency from Baseline to the Maintenance Period.
Time Frame: 8-week Baseline Period (Visit 1 to 3) and 12-week Maintenance Period (Visit 5 to 8)
Population: The Full Analysis Set consists of all subjects who were randomized, received at least 1 dose of study drug, and had at least 1 post-baseline efficacy assessment.
Measure: Median (Full Range); unit: Seizures per 28 days
Arm/Group | Placebo | Lacosamide 200 mg/Day | Lacosamide 400 mg/Day
Number analyzed (Participants) | 183 | 182 | 179
Seizures per 28 days | -1.22 [-93.0 to 39.8] | -3.33 [-754.3 to 165.2] | -4.50 [-97.5 to 28.2]
Statistical Analysis 1: Comparison: Placebo vs Lacosamide 400 mg/Day; To avoid inflation of Type I error, hypothesis testing followed predefined hierarchical procedure starting LCM 400 mg/day treatment group versus the placebo group. If the test was not statistically significant, the procedure stopped and no Groups were declared different from placebo. If the test was statistically significant, the treatment group was considered different from placebo and the procedure continued with the LCM 200 mg/day treatment group; Test type: Superiority or Other; p < 0.001, ANCOVA — Significant at the 0.05 level. This testing procedure is considered a closed testing procedure and no adjustment of the significance level was necessary; % Reduction over Placebo = 39.6, 95% CI 2-sided [30.5 to 47.6]
Statistical Analysis 2: Comparison: Placebo vs Lacosamide 200 mg/Day; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; % Reduction over Placebo = 29.4, 95% CI 2-sided [18.7 to 38.7]

2. Secondary Outcome: The Proportion of Individual Patients Who Experience a 50 % or Greater Reduction in Seizure Frequency From Baseline to the Maintenance Period (50 % Responder Rate)
Time Frame: 8-week Baseline Period (Visit 1 to 3) to the 12-week Maintenance Period (Visit 5 to 8)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Lacosamide 200 mg/Day | Lacosamide 400 mg/Day
Number analyzed (Participants) | 183 | 182 | 179
participants | 36 | 70 | 88

3. Secondary Outcome: Percent Change in Partial-Onset Seizure Frequency Per 28 Days From Baseline to the Maintenance Period
Description: Calculates as 28-day seizure frequency during the Maintenance Period - 28-day seizure frequency during the Baseline Period, divided by the 28-day seizure frequency during the Baseline Period with this quantity multiplied by 100. A negative value in percent change from Baseline indicates a decrease in Partial-Onset Seizure frequency from Baseline to the Maintenance Period.
Time Frame: 8-week Baseline Period (Visit 1 to 3) to the 12-week Maintenance Period (Visit 5 to 8)
Population: as for outcome 1
Measure: Median (Full Range); unit: percentage change
Arm/Group | Placebo | Lacosamide 200 mg/Day | Lacosamide 400 mg/Day
Number analyzed (Participants) | 183 | 182 | 179
percentage change | -10.10 [-97.6 to 233.5] | -36.75 [-100.0 to 185.5] | -48.78 [-100.0 to 346.4]

4. Secondary Outcome: Change in Partial-Onset Seizure Frequency Per 28 Days From Baseline to the Treatment Period (i.e., Titration + Maintenance Period)
Description: Partial-onset seizure (POS) frequency per 28 days was calculated as:
  POS frequency = (Number of POS over the specified time interval) / (Number of days in the interval with available diary data) x 28.
  A negative value in Change in Partial-onset seizure frequency indicates a reduction of Partial-onset seizure frequency from Baseline to the Treatment Period.
Time Frame: 8-week Baseline Period (Visit 1 to 3) to the 16-week Treatment Period (Visit 3 to 8)
Population: as for outcome 1
Measure: Median (Full Range); unit: Seizures per 28 days
Arm/Group | Placebo | Lacosamide 200 mg/Day | Lacosamide 400 mg/Day
Number analyzed (Participants) | 183 | 182 | 179
Seizures per 28 days | -1.10 [-102.4 to 102.5] | -3.39 [-670.0 to 138.9] | -4.00 [-92.4 to 34.2]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from Baseline to the end of the study (up to Week 19).
Description: Treatment Emergent Adverse Events (TEAEs) refer to the Safety Set (SS). The SS includes all randomized subjects who took at least 1 dose of study drug.
Arm/Group | Placebo | Lacosamide 200 mg/Day | Lacosamide 400 mg/Day
Serious Adverse Events (participants affected / at risk) | 4/184 | 2/183 | 9/180
Other Adverse Events (participants affected / at risk) | 77/184 | 87/183 | 112/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=184) | Lacosamide 200 mg/Day (N=183) | Lacosamide 400 mg/Day (N=180)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Epileptic psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=184) | Lacosamide 200 mg/Day (N=183) | Lacosamide 400 mg/Day (N=180)
Diplopia (Eye disorders) | 4 (5) | 4 (8) | 13 (15)
Vomiting (Gastrointestinal disorders) | 4 (4) | 5 (6) | 14 (18)
Nausea (Gastrointestinal disorders) | 9 (10) | 7 (8) | 10 (11)
Nasopharyngitis (Infections and infestations) | 24 (41) | 28 (40) | 29 (36)
Upper respiratory tract infection (Infections and infestations) | 22 (31) | 10 (14) | 19 (28)
White blood cell count decreased (Investigations) | 2 (2) | 8 (14) | 10 (12)
Dizziness (Nervous system disorders) | 24 (32) | 33 (57) | 63 (118)
Somnolence (Nervous system disorders) | 9 (10) | 18 (26) | 19 (21)
Headache (Nervous system disorders) | 11 (21) | 16 (18) | 19 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days